CLINICAL TRIAL: NCT03388021
Title: Routine Versus Selective Completion Angiography After Thromboembolectomy in the Treatment of Acute Lower Limb Ischemia: A Randomized Controlled Trial
Brief Title: A Trial Comparing Routine Versus Selective Use of Completion Angiography After Surgical Thromboembolectomy in the Treatment of Acute Lower Limb Ischemia and Their Impacts on Limb Salvage Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Elshafie, Assistant Lecturer of vascular surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD/85
Record Dates: First submitted 2017-12-23; First posted 2018-01-02 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Acute Limb Ischemia
Keywords: limb ischemia; completion angiography; thromboembolectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine use of completion angiography after thromboembolectomy (Experimental): this group will undergo surgical revascularization followed by routine completion angiography assisted with one of these adjuvant techniques as:
  1. Thromboembolectomy under fluoroscopic guidance using Fogarty over the wire
  2. Balloon angioplasty and/or stenting
  3. Intraarterial thrombolysis
  Aiming to correct any residual angiographic lesion as:
  1. Residual thrombus
  2. Retained embolus
  3. Atheromatous plaque
  Interventions: Procedure: completion angiography followed by endovascular treatment of residual or underlying lesions
- if the results were not satisfactory intraoperatively as fail (Active Comparator): this group will undergo surgical thromboembolectomy. if the results were not satisfactory intraoperatively as failure to advance the Fogarty catheter or to get satisfactory inflow or backflow or Extraction of intimal fragments.patient will undergo diagnostic angiography and endovascular or surgical intervention according to result of diagnostic angiography.
  Interventions: Procedure: completion angiography followed by endovascular treatment of residual or underlying lesions

INTERVENTIONS:
Procedure: completion angiography followed by endovascular treatment of residual or underlying lesions — completion angiography followed by endovascular treatment as thromboembolectomy under fluoroscopic guidance using Fogarty over the wire, angioplasty, stenting, or Intraarterial thrombolysis to treat residual or underlying lesions

SUMMARY:
this randomized controlled trial will compare the impact of routine use of completion angiography versus using it on selective bases after thromboembolectomy in patients with acute lower limb ischemia and their impact on limb salvage rates

ELIGIBILITY:
Inclusion Criteria:

* Grade I (1) (viable) acute ischemia which there is no immediate threat of limb loss; the patient is presented with neither sensory nor motor weakness and there are audible Doppler signals in both arteries and veins.
* Grade IIA (2 A) (marginally threatened) acute ischemia which needs proper treatment to save the limb; the patient is presented with a minimal sensory loss, no motor weakness, inaudible arterial Doppler signals but the venous Doppler signals are still audible.
* Grade IIB (2 B) (immediately threatened) acute ischemia which needs immediate revascularization to save the limb; the patient is presented with a sensory loss associated with rest pain, mild to moderate motor weakness, inaudible arterial Doppler signals but the venous Doppler signals are still audible.

Exclusion Criteria:

* Traumatic or iatrogenic acute limb ischemia
* Grade III acute ischemia (irreversible) with major tissue loss and major amputation is inevitable; the patient presented with sensory and motor loss, inaudible arterial and venous Doppler signals.
* Patients With occluded bypass graft.
* Acute limb ischemia due to intra-arterial injection
* Patients with chronic renal impairment (serum creatinine > 1.2) or with a history of contrast-induced nephropathy.
* Acute lower limb ischemia due to thrombosed aneurysms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-02-04 (Actual); Study Completion 2018-02-04 (Actual)

PRIMARY OUTCOMES:
limb salvage rate | 2 years after operation
  free from major amputation
primary patency | 2 years after operation
  free from reintervention
mortality rate | 30 days after operation
  death related from the intervention

SECONDARY OUTCOMES:
complication rates | 2 years after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Al Dakhlia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutherford RB. Clinical staging of acute limb ischemia as the basis for choice of revascularization method: when and how to intervene. Semin Vasc Surg. 2009 Mar;22(1):5-9. doi: 10.1053/j.semvascsurg.2008.12.003. PMID 19298929
- [Background] Ouriel K. Endovascular techniques in the treatment of acute limb ischemia: thrombolytic agents, trials, and percutaneous mechanical thrombectomy techniques. Semin Vasc Surg. 2003 Dec;16(4):270-9. doi: 10.1053/j.semvascsurg.2003.08.004. PMID 14691769
- [Result] Zaraca F, Stringari C, Ebner JA, Ebner H. Routine versus selective use of intraoperative angiography during thromboembolectomy for acute lower limb ischemia: analysis of outcomes. Ann Vasc Surg. 2010 Jul;24(5):621-7. doi: 10.1016/j.avsg.2009.12.006. Epub 2010 Apr 2. PMID 20363108
- [Result] Zaraca F, Ponzoni A, Sbraga P, Stringari C, Ebner JA, Ebner H. Does routine completion angiogram during embolectomy for acute upper-limb ischemia improve outcomes? Ann Vasc Surg. 2012 Nov;26(8):1064-70. doi: 10.1016/j.avsg.2011.12.012. Epub 2012 Jun 26. PMID 22743219
- [Result] de Donato G, Setacci F, Sirignano P, Galzerano G, Massaroni R, Setacci C. The combination of surgical embolectomy and endovascular techniques may improve outcomes of patients with acute lower limb ischemia. J Vasc Surg. 2014 Mar;59(3):729-36. doi: 10.1016/j.jvs.2013.09.016. Epub 2013 Dec 15. PMID 24342067
- [Result] Argyriou C, Georgakarakos E, Georgiadis GS, Antoniou GA, Schoretsanitis N, Lazarides M. Hybrid revascularization procedures in acute limb ischemia. Ann Vasc Surg. 2014 Aug;28(6):1456-62. doi: 10.1016/j.avsg.2014.01.019. Epub 2014 Feb 11. PMID 24530573